CLINICAL TRIAL: NCT06806449
Title: Results of Silver-coated Resection Prostheses in the Two-stage Treatment of Periprosthetic Knee Infections with Bone Deficiency
Brief Title: Results of Silver-coated Resection Prostheses in the Treatment of Periprosthetic Knee Infections with Bone Deficiency
Acronym: MEGAPJI
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: MEGAPJI
Record Dates: First submitted 2024-12-01; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-12

CONDITIONS: PJI
Keywords: two-stage treatment; PJI; silver-coated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to evaluate the infection control and mid-term survival of silver-coated articulated megaprosthetic and knee arthrodesis implants in PJI patients with bone stock deficiency and treated with two-stage protocol.

DETAILED DESCRIPTION:
The majority of studies investigating the outcomes of silver-coated megaprostheses have evaluated case histories of megaprostheses in oncologic patients, while there is little evidence in the Literature of the outcomes of silver-coated megaprostheses in the treatment of infections in non-oncologic patients.

Knowing the mid- to long-term results of this type of implant is of great importance to inform the patient regarding expectations after surgery.

Obtaining more results and data on the treatment of knee PJI with silver-coated megaprostheses could pave the way for the design of prospective randomized comparative trials aimed at establishing the gold standard of treatment.

It is a nonprofit, observational, cohort, retrospective and prospective, multicenter, national study. Patients will be treated according to clinical practice in accordance with the judgment of the clinician.

The biographical and clinical-radiographic data that will be collected are:

1. Pre-operative data: timing of infection, bacterial population involved, primary or revision implant (specifying number and type of surgeries and in case of use of implants, number and type of implants), baseline characteristics of the patient (sex, age, date of previous surgeries, number and type of previous surgeries, comorbidities, ASA score, smoking, alcohol, etc.), local knee problems, investigations performed.
2. Intra-operative data: The surgical technique will be described with reference to type of access, procedure, type of resection (distal femoral, proximal tibial, both) and length of resection, type of spacer used, sizes of prosthetic components implanted and prosthetic model, possible use of cementation or grafts (specifying nature of graft), possible occurrence of intraoperative complications.
3. Postoperative data: antibiotic therapy, results of histological and culture investigations, postoperative complications, implant status at follow-up (specifying in case of failure, the cause of failure), duration of follow-up.

All data and clinical and radiographic material will be collected together and analyzed at IRCCS Azienda Ospedaliero Universitaria di Bologna. All radiographic measurements will be performed by 3 independent operators after evaluation of intra- and inter-observer reliability on 10 random patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of periprosthetic knee infection on primary or already revised implants
* Treatment of infection with two-stage protocol
* Placement of articulated knee megaprosthesis (distal femoral or proximal tibial resection) or arthrodesis, silver-coated.
* Clinical and radiographic follow-up obtained or obtainable greater than or equal to 24 months.
* Completeness of clinical-radiographic documentation
* Obtainment of informed consent
* Age>=18 years

Exclusion Criteria:

* Unfit patients
* Patient with a history of oncology
* Patient with contraindications to taking radiographs at follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at the Orthopedics and Traumatology Operating Unit of IRCCS Azienda Ospedaliero Universitaria di Bologna, Policlinico di S.Orsola and other national centers between January 2020 and December 2024 with silver-coated knee megaprosthesis in the two-stage treatment of knee PJI.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2023-08-20 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
Infection status | through study completion, an average of 1 year
  absence of clinical radiological and/or laboratory signs of infection or infected.

SECONDARY OUTCOMES:
Incidence of complications unrelated to prosthesis infection in the two different stages of the protocol, also analyzing the number of "first stage" repetitions | Within 8 weeks and 24 months
  Number and type of non-infection-related complications of "first-stage" within 8 weeks and "second-stage" within 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Sambri, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (3):
- Italy (3):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna
  - Azienda Ospedaliero Universitaria Careggi, Florence, Florence
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Pisa